CLINICAL TRIAL: NCT03189043
Title: Controlled Crossover Study of AIONX Antimicrobial Surface for the Prevention of Healthcare-associated Infections
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aionx, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Jose Stoute, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 7371
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Healthcare Associated Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Use of antimicrobial surface
  Interventions: Device: Antimicrobial Surface
- Control (No Intervention): No antimicrobial surface

INTERVENTIONS:
Device: Antimicrobial Surface — Antimicrobial Surface
  Arms: Test

SUMMARY:
This is a controlled open label efficacy study of Aionx antimicrobial surface for the prevention of healthcare-associated infections.

DETAILED DESCRIPTION:
The study is an open label controlled efficacy trial of Aionx patented antimicrobial surface for the prevention of healthcare-associated infections (HAIs). It will take place at Penn State Hershey. Half of the single occupancy rooms of the 5th and 7th floor will be assigned to contain the antimicrobial surface at five locations: bed rails, overbed table, door handles, counter, and arm rests of bedside chair. The remaining rooms will serve as controls. Data on HAIs will be gathered for all the patients admitted to the rooms during the duration of the study. After 45 days the rooms will be flipped so that test rooms become controls and control rooms become test rooms. The duration of the study will be for a minimum of 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a single occupancy room in a participating floor at Hershey Medical Center

Exclusion Criteria:

* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Healthcare-Associated Infections | 90 days
  Healthcare-Associated Infections

SECONDARY OUTCOMES:
30-day Readmission for infection | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Stoute, M.D., Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No